CLINICAL TRIAL: NCT06102850
Title: Adaptation of Critical Time Intervention for Young Adults With Mental Health Challenges in the Transition From Homelessness to Housing
Brief Title: Adaptation of Critical Time Intervention for Young Adults With MH Challenges
Acronym: CTI-YAMH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Sarah C Narendorf, Associate Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R34MH129542-01A1 (NIH)
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: This study includes a phased open trial, first using a single group feasibility pilot (n=8) to refine the intervention manuals, then employed a randomized parallel feasibility pilot (n=26 in each group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Condition, CTI-YAMH (Experimental): Participants receive the CTI-YAMH intervention in conjunction with rapid rehousing supports for the 6 month intervention
  Interventions: Behavioral: Critical Time Intervention for Young Adults with Mental Health conditions
- Treatment as Usual Condition (No Intervention): Participants will be assigned to a housing program at another agency that provides rapid rehousing with usual supports

INTERVENTIONS:
Behavioral: Critical Time Intervention for Young Adults with Mental Health conditions — SIx month supportive intervention involving CTI phased based casemanagement, support from a peer support specialist, and support from a mental health liaison
  Arms: Intervention Condition, CTI-YAMH

SUMMARY:
Young adults experiencing homelessness have high rates of mental health conditions but low rates of service utilization and the point of transition from homelessness to supported housing provides a window of opportunity for intervention. The goal of this study is to adapt the evidenced-based intervention, Critical Time Intervention, for young adults with mental health conditions who are entering a rapid rehousing program and test the adapted intervention in a randomized feasibility pilot trial. Participants in the pilot trial will be asked to participate in the CTI-YAMH intervention that involves structured case management and supports from a mental health liaison and a peer support specialist. After a pilot feasibility phase (n=8), we will test the intervention by randomly assigning young adults on the housing wait list to a housing program with CTI-YAMH (n=26) or to get housing supports from another agency that does not provide CTI-YAMH (treatment as usual, n=26).

DETAILED DESCRIPTION:
The design of the phased open trial allows for us to test and further refine our intervention procedures, then include this learning in a randomized feasibility pilot. This will enable us to examine several issues that we anticipate will need refinement prior to larger testing in a fully powered future large study. Our sample (n=60) will include young adults (age 18-24) who have qualified for RRH supports. Entry into the homelessness system is managed through a coordinated access system with a consistent assessment process and centralized wait list which is prioritized based on a screener that asks respondents to self-report whether they have been diagnosed with a mental disorder. Young adults are assigned to a RRH case manager based on capacity across agencies that provide RRH including Covenant House TExas (CHT). CTI-YAMH targets young adults with mental health symptoms and will be implemented at CHT. The screening tool used to prioritize assignment to housing asks for a self-report of mental health symptoms as well as other risk factors that give a housing priority score. When CHT has capacity for a new youth, we will work with the coordinated access system to match and enroll two young adults with similar priority scores into our study after screening for mental health symptoms, then randomize one to CHT and one to another agency providing young adult RRH with capacity (TAU). We will closely track the feasibility of this real-world process, keeping track of the number of YAEH who are on the waiting list, number contacted, number successfully enrolled, and number that meet our enrollment criteria. For this study, we will partner with CHT which currently employs three RRH case managers who each carry a caseload of 18 young adults.

For the first phase of the open trial, we aim to recruit and enroll a sample of 8 participants. We anticipate this will take approximately 3 months which will enable us to refine our enrollment procedures and finalize intervention procedures. After 6 months we will move into the next phase. For the second phase of the open trial, we aim to recruit a sample of 52 young adults, 26 for each condition over the course of the 12-month period. Across the community, the average length of stay in RRH is 12 months so without accounting for likely expansion, we anticipate that there will be approximately 4-5 intakes per month for the CHT RRH program at current size. Given the new focus on young adults in the community and potential expansion of RRH services at CHT, we expect that this number will increase as services ramp up. Based on our prior research, we estimate that 60-75% will screen positive for mental health problems as assessed with the Kessler-6 so at current capacity we would identify 3-4 participants per month that are eligible for the study and enroll 2-3 of these for approximately 12 months in the intervention condition and 2-3 participants per month for 12 months in the TAU condition..condition.

Enrollment and Data Collection Procedures. For both phases, young adults (age 18-24) on the housing eligibility list will be screened for study criteria (meeting criteria for psychological distress on Kessler-6 [74] or self-reported prior diagnosis of depression, anxiety, bipolar or a psychotic disorder with ongoing symptoms) and invited to participate at the point of assignment to RRH. Young adults will be told of the opportunity to participate in the study at the time of eligibility assessment for housing and asked for permission to provide their names to the study team if interested. For the first phase we will attempt to enroll all those assigned to RRH at CHT who meet our criteria. For the second phase, when housing is about to be assigned for CHT, we will attempt to enroll two similar young people and assign one to CHT and one to TAU. For both phases 1 and 2, we will contact young people about their interest, then schedule a baseline interview to be held over zoom or by phone lasting approximately one hour. Interviewers will obtain informed consent electronically signed through DocuSign and administer the survey via phone or zoom with each meeting lasting approximately one hour. This format enables us to be flexible and responsive in scheduling interviews. If participants do not have access to a phone or zoom, researchers have the ability to meet clients in the agency where they individual is connected to a case manager. In order to track outcomes through the course of the 6-month intervention, research assistants we will administer surveys at baseline, the midpoint (3 months), end of the intervention (6 months) and 6 month6-month follow-up (12 months). Survey data at each measurement point will be collected on tablets using a questionnaire programmed in Qualtrics. For those in phase 1, we will also conduct qualitative interviews (n=8) and will also interview each of the professionals involved in implementing it (n=5) to explore qualitatively how the intervention activities hit the hypothesized targets of the intervention and allow the potential for other key mechanisms to emerge as well as assess implementation outcomes of acceptability and appropriateness. Qualitative interviews will be conducted using a semi-structured interview guide and will be digitally recorded, then transcribed. If participants do not want to be recorded, detailed notes will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Young adults (age 18-24) on the housing eligibility list assigned to rapid rehousing
* Positive for psychological distress on Kessler-6 or self-reported prior diagnosis of depression, anxiety, bipolar or a psychotic disorder with ongoing symptoms

Exclusion Criteria:

* Age 25 or older
* Not English speaking
* No eligible for rapid rehousing based on housing priority score

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Housing Stability | Baseline, 3 mo, 6 mo, 12 mo
  Housing Security Scale Number of days homeless, Number of moves in prior 90 days
Mental Disorder | Baseline, 12 mo.
  Diagnosis of Common Disorders i.e. Depression, Anxiety, Bipolar, Psychotic Disorders
Depressive Symptoms | Baseline, 3 mo, 6mo, 12 mo.
  PHQ-9
Anxiety Symptoms | Baseline, 3 mo, 6mo, 12 mo.
  GAD-7
PTSD Symptoms | Baseline, 3 mo, 6mo, 12 mo.
  Primary Care PTSD Screen

SECONDARY OUTCOMES:
Treatment Engagement | Baseline, 3 mo, 6mo, 12 mo.
  Self-report of taking medication, attending appointments;
  Client Engagement in Child Protective Services Scale, modified for mental health services

CONTACTS AND LOCATIONS:
Locations (1):
- Covenant House Texas, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded to the NIMH NDA using GUID identifiers
Supporting Information: Study Protocol, ICF
Time Frame: in accordance with data sharing requirements for NIMH
Access Criteria: Institutional level through the NDA
URL: https://nda.nih.gov/

REFERENCES:
- [Derived] Narendorf SC, Munson MR, Khan U, Brown M, Gomez G, Santa Maria D, Gilmer T, Gattis MN, Hayward P, Herman D. Study protocol for a feasibility evaluation of Charge Up!: an adaptation of Critical Time Intervention for young adults moving from homelessness to housing. Pilot Feasibility Stud. 2025 Jul 2;11(1):91. doi: 10.1186/s40814-025-01677-7. PMID 40605122